CLINICAL TRIAL: NCT00003558
Title: A Randomized Phase III Trial of Paclitaxel, Carboplatin and Etoposide Vs. 5-Fluorouracil and Folinic Acid in the Treatment of Patients With Adenocarcinoma of Unknown Primary Site
Brief Title: Chemotherapy in Treating Patients With Cancer of Unknown Primary Origin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: DUT-KWF-CKVO-9801; CDR0000066622 (Registry Identifier: PDQ (Physician Data Query)); EU-98023
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2003-02

CONDITIONS: Carcinoma of Unknown Primary
Keywords: adenocarcinoma of unknown primary; newly diagnosed carcinoma of unknown primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Carboplatin; Etoposide; Fluorouracil; Leucovorin; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: etoposide
Drug: fluorouracil
Drug: leucovorin calcium
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective for cancer of unknown primary origin.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different regimens of combination chemotherapy in treating patients with cancer of unknown primary origin.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival after treatment with paclitaxel, carboplatin, and etoposide and after treatment with fluorouracil and leucovorin calcium in patients with adenocarcinoma of unknown primary.
* Compare the response rates, progression free survival, toxicity profile, and quality of life between the two regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center and presence or absence of liver metastases.

Patients are randomly assigned to one of two treatment arms.

* Arm I: Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1, and oral etoposide on days 1-10. Treatment is repeated every 3 weeks for up to four courses.
* Arm II: Patients receive leucovorin calcium IV over 2 hours followed by fluorouracil IV over 24 hours weekly for 6 weeks. Treatment is repeated every 7 weeks for up to two courses.

Patients are followed every 3 months after treatment for 1 year or until death. Quality of life questionnaires are completed at each follow-up.

PROJECTED ACCRUAL: Approximately 120-140 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of any differentiation grade

  * Excludes the following "treatable" conditions:

    * Axillary node involvement
    * Peritonitis carcinomatosis
    * Blastic bone metastases and/or elevated PSA
    * Squamous cell cancer with cervical or inguinal presentation
    * Poorly differentiated carcinoma

      * Neuroendocrine tumors OR
      * Tumors located in the mediastinum, retroperitoneum, or nodes
* At least one measurable metastatic site
* No brain or meningeal metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Hematopoietic:

* Leukocyte count at least 4,000/mm3
* Thrombocyte count at least 100,000/mm3

Hepatic:

* Bilirubin less than 1.4 mg/dL
* AST and ALT less than 3 times upper limit of normal
* No cirrhosis of the liver

Renal:

* Creatinine less than 1.7 mg/dL

Cardiovascular:

* At least 3 months since myocardial infarction
* No congestive heart failure, tachydysrhythmia, or unstable angina pectoris

Other:

* Not pregnant or nursing
* Negative pregnancy test
* No active infection
* No other serious illness or medical condition
* No current or prior malignancy except nonmelanomatous skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy (no greater than 25% of bone marrow)

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 1998-08

CONTACTS AND LOCATIONS:
Overall Officials: R. L. Jansen, MD, PhD, Study Chair — Academisch Ziekenhuis Maastricht
Locations (2):
- Netherlands (2):
  - Academisch Ziekenhuis Maastricht, Maastricht
  - St. Elisabeth Ziekenhuis, Tilburg